CLINICAL TRIAL: NCT06746766
Title: Registry Study on Rare Cancers in Korea
Acronym: rarecancer
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, Principal Investigator, Yonsei University
Other Study IDs: 4-2024-1207; 4-2024-1207 (Other: Severance Hospital, IRB)
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Rare Cancer
Keywords: Rare Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the participation rate of patients with registered rare cancers in clinical research.

DETAILED DESCRIPTION:
Data collection includes:

* Clinical characteristics (diagnosis, treatment information, primary/metastatic sites, staging, gender/age)
* Survival information (diagnosis date, recurrence date, death date, disease progression)
* Pathological information (diagnosis, genomic information)

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years
* Confirmed rare cancer
* Life expectancy ≥3 months

Exclusion Criteria:

-Serious or unstable medical/psychiatric conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data collection includes:
  * Clinical characteristics (diagnosis, treatment information, primary/metastatic sites, staging, gender/age)
  * Survival information (diagnosis date, recurrence date, death date, disease progression)
  * Pathological information (diagnosis, genomic information)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Establish a registry | 1 year
  Establish a registry of rare cancer patients visiting the institution

SECONDARY OUTCOMES:
Clinical trial registration rate (%) | 1 year
  Clinical trial registration rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Song Kim, MD, Ph.D, Principal Investigator — Yonsei Cencer center
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Gatta G, Capocaccia R, Trama A, Martinez-Garcia C; RARECARE Working Group. The burden of rare cancers in Europe. Adv Exp Med Biol. 2010;686:285-303. doi: 10.1007/978-90-481-9485-8_17. PMID 20824452
- [Background] Very rare cancers--a problem neglected. Lancet Oncol. 2001 Apr;2(4):189. doi: 10.1016/s1470-2045(00)00273-4. No abstract available. PMID 11905758
- [Background] Pritchard-Jones K, Kaatsch P, Steliarova-Foucher E, Stiller CA, Coebergh JW. Cancer in children and adolescents in Europe: developments over 20 years and future challenges. Eur J Cancer. 2006 Sep;42(13):2183-90. doi: 10.1016/j.ejca.2006.06.006. PMID 16919780